CLINICAL TRIAL: NCT06285266
Title: Investigation of Nursing Students' Perceptions of the Clinical Learning Environment in Surgical Services and Their Participation in Clinical Practices: A Cross-Sectional Study
Brief Title: Nursing Students' Perceptions and Participation in Surgical Clinical Learning
Acronym: NSPSCP_CL
Status: Not yet recruiting | Type: Observational
Sponsor: Kilis 7 Aralik University (Other)
Collaborators: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, İslam Elagöz, PhD, Kilis 7 Aralik University
Other Study IDs: kilis_1
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Clinical Practice
Keywords: Nursing Student; Surgical Services; Clinical Practice; Clinical Learning Environment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This cross-sectional study investigates the perceptions of nursing students regarding the clinical learning environment (CLE) in surgical services and their participation in clinical practices. Surgical services present a complex, dynamic, and intense learning environment crucial for the development of nursing students' professional competencies. The study explores the challenges nursing students face in these settings, including limited opportunities for participation in intraoperative processes and intensive care units, and the impact of these challenges on their learning outcomes and professional development.

Previous research has highlighted various factors that can either facilitate or hinder nursing students' ability to engage effectively in clinical practices, such as the learning atmosphere, support from nurse educators, peer support, and effective communication. However, there is a noted gap in understanding the specific difficulties encountered in surgical services, the adequacy of students' clinical skills and knowledge, and their ability to apply theoretical knowledge in practice.

By examining nursing students' experiences, this study aims to shed light on the suitability and quality of CLEs in surgical services, contributing valuable insights for optimizing clinical learning and enhancing nursing education programs. The hypotheses tested whether nursing students' perceptions of CLEs in surgical services and their participation in clinical practices are influenced by their descriptive characteristics.

Keywords: Nursing Student, Surgical Services, Clinical Practice, Clinical Learning Environment

DETAILED DESCRIPTION:
INTRODUCTION Surgical Services provide a critical, complex, dynamic, and intense Clinical Learning Environment (CLE) for Nursing Students (NS) to learn (Namara CM 2023) (Atkinson RB 2023). The instantaneous changes in the conditions of patients in surgical services, measures to prevent infection due to incision, and the management of symptoms related to surgery require a professional approach (Engel JS 2023). Especially, participation of NS in clinical practices during the intraoperative process and in the intensive care unit is often not possible (Numara RB 2023). The quality of CLEs in surgical services raises doubts about students' learning outcomes. Numerous studies suggest that not all clinical settings are conducive to learning (Chan A 2018) (Lee T 2023) (Kalyani MN 2019) (Günay U 2018).

Nursing is an applied science. For professional competence, the integration of theoretical and practical knowledge is required (Carless-Kare S.2023). The suitability of CLEs allows Nursing Students (NS) to perform and learn basic nursing practices. Nursing practices develop NS's psychomotor, cognitive, affective skills, as well as their resilience (Saka K 2023). This development depends on the diversity of practices, frequency of practice, and being in a real clinical environment (Karadağ et al., 2013). Practices in clinical settings enable NS to observe, take responsibility, learn to act according to the patient's clinical condition, make clinical decisions, and learn to work as a member of the health team (Karadağ et al., 2013). NS are expected to participate in nursing practices in clinical settings to enrich their experiences and practice development (Amsalu et al., 2020). However, it is reported that NS face difficulties in the clinical area and cannot always participate sufficiently in clinical practices (Kalyani MN 2019) (Günay U 2018) (Yazdankhahfard, M 2020) (Carless-Kane S 2023) (Günay U 2018). A qualitative study reported that NS find their clinical knowledge and skills insufficient and cannot transfer theoretical knowledge into practice (Günay U 2018).

BACKGROUND Previous studies have determined the levels and frequencies at which nursing students perform basic nursing practices (Lee T 2023) (Amsalu et al., 2020) (Carless- Kane S-2023) (Günay U 2018) (Kalyani MN 2019).

The findings of these studies have revealed many factors that could either hinder or facilitate nursing students' ability to practice and gain proficiency in clinical practice areas (Carless-Kane S 2023) (Günay U 2018) (Kalyani MN 2019). A conducive clinical atmosphere for learning (Kalyani MN 2019), supportive attitudes of nurse educators towards students (Günay U 2018), peer support in the clinical environment (Carless-Kane S 2023), and effective communication (Günay U 2018) have been determined to be associated with clinical practice proficiency. The presence of too many students in the practice area (Arkan 2018), insufficient number of patients (Arkan 2018) (Amsalu 2020), and lack of teaching staff (Günay U 2018) (Arkan 2018) (Amsalu 2020) have been shown to decrease clinical practice proficiency.

Previous studies have been conducted to determine the suitability, quality, and student satisfaction of CLEs (Saka K 2023) (Yazdankhahfard M 2020) (Lee T 2023) (Atkinson RB 2023) (Namara CM 2023). However, the challenges NS face in CLEs in surgical services, their opportunities to participate in practices, and the impact of these experiences on students' professional development have not yet been fully understood. Studies addressing the challenges faced by nursing students in surgical services, strategies to overcome these challenges, and their participation status in practices should be conducted. The findings could significantly contribute to optimizing clinical learning in surgical services in nursing education programs and enhancing students' effectiveness in these environments. This study was conducted with the aim of determining the perceptions of nursing students regarding clinical learning environments and their participation in clinical practices in surgical services.

The following hypotheses were tested in this study:

H0: Nursing students; perceptions of clinical learning environments in surgical services, their participation status, and descriptive characteristics are not affected.

H1: Nursing students; perceptions of clinical learning environments in surgical services, their participation status, and descriptive characteristics are affected.

ELIGIBILITY:
Inclusion Criteria:

* Nursing students taking a surgical course for the first time,
* Those who are not graduates of a vocational health high school,
* Those not working as health professionals,
* Nursing students willing to participate in the study were included.

Exclusion Criteria:

* Students who wished to withdraw from the sample at any stage of the research were excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of nursing students enrolled in a surgical nursing course for the first time, excluding those with a vocational health high school background or current healthcare professionals. This selection aims to ensure participants have similar educational experiences and are in a critical phase of integrating theoretical knowledge with practical skills. Focusing on students not yet working in health services allows for a clearer assessment of educational impacts without professional biases. Participation is voluntary, emphasizing engaged learners likely to provide insightful feedback on their clinical learning environment in surgical settings. This approach aims to identify educational facilitators and barriers within a specific, challenging clinical context.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Descriptive Characteristics Form | up to 18 weeks
  The Descriptive Characteristics Form includes questions aimed at determining students' age, gender, high school from which they graduated, and their perceptions regarding the adequacy of their participation in clinical practices in surgical services.
Clinical Learning Environment Scale (CLES): | up to 18 weeks
  The scale was developed by Dunn and Burnett in 1995 (Dunn & Burnett, 1995) and was adapted into Turkish by Sarı in 2001 (Sarı, 2001). The scale consists of 22 items across 5 sub-dimensions: "Staff-Student Relationships" (items 7, 8, 15, 19, 20, and 21), "Roles of Teaching Staff" (items 3, 5, 11, and 12), "Patient Relationships" (items 2, 10, 14, and 22), "Student Satisfaction" (items 9, 16, 17, and 18), and "Hierarchy and Routines" (items 1, 4, 6, and 13). The lowest possible score on the scale is 22, and the highest is 110, with higher scores indicating a more positive evaluation of the clinical learning environment. The original scale's Cronbach's alpha reliability coefficient was calculated as and the Turkish adaptation's Cronbach's alpha reliability coefficient was calculated as The Cronbach's alpha reliability coefficient for this study was calculated as
Clinical Practice Participation Determination Form: | up to 18 weeks
  The Clinical Practice Participation Determination Form was created by the researchers following a review of sources. It contains 30 multiple-choice questions aimed at determining nursing students' ability to participate in clinical practices. To establish the form's content validity, expert opinions were obtained from 5 nursing academics. The Content Validity Index (CVI) was calculated to be 0.98, and the form was deemed suitable for the research. Since the CVI is 0.98 > 0.80, it was decided that the data collection forms are appropriate for this research (Davis and Grant, 1993). The Cronbach's alpha reliability coefficient for the Clinical Practice Participation Determination Form was calculated as Clinical Practice Participation Facilitators and Barriers The Content Validity Index (CVI) was calculated to be 0.98, and the form was deemed suitable for the research.

CONTACTS AND LOCATIONS:
Overall Officials: islam elagöz, MsC, Study Chair — devlet hastanesi

IPD SHARING:
Plan to Share IPD: No
Yes, there is a plan to make individual participant data (IPD) available to other researchers. This will include de-identified participant data that underpinned the study's findings, such as responses to surveys or questionnaires, clinical practice participation details, and any additional collected metrics relevant to the study's objectives. Access to this data will be provided upon reasonable request to the principal investigator, following the completion of the study and publication of its primary outcomes. The data sharing plan is designed to ensure that participant confidentiality is maintained, in compliance with ethical guidelines and regulations governing research data. Researchers interested in accessing the IPD will be required to submit a proposal outlining their intended use of the data, which will be reviewed for alignment with the original study's ethical approval and objectives.